# UNIVERSITY OF WASHINGTON CONSENT FORM

# Effects of Isotretinoin on CYP2D6 Activity

#### **Researchers:**

# **Lead Researcher and Contact Person for Subjects:**

Mary F. Hebert, PharmD, FCCP Professor Pharmacy 206-616-5016

**Coordinator:** 

Alicia Stark Student Res. Assist. Pharmacy (360) 921-3715

24-hour emergency telephone number: 206-598-6190 (Paging Operator), ask for Dr. Vary.

## Researchers' statement

Throughout this form we refer to 'you' as the subject. If you are providing permission for a minor to participate, 'you' refers to 'your child'. We are asking you to be in a research study. The purpose of this consent form is to give you the information you will need to help you decide whether to be in the study or not. Please read the form carefully. You may ask questions about the purpose of the research, what we would ask you to do, the possible risks and benefits, your rights as a volunteer, and anything else about the research or this form that is not clear. When we have answered all your questions, you can decide if you want to be in the study or not. This process is called "informed consent." We will give you a copy of this form for your records.

## **PURPOSE OF THE STUDY**

Research tells us that chemicals like vitamin A are involved in determining how the body handles drugs. The purpose of this work is to see if isotretinoin, an acne medication similar to vitamin A, changes how the body handles dextromethorphan, a cough medication. This study will include 50 patients that will be receiving isotretinoin for clinical reasons.

### STUDY PROCEDURES

If you agree to participate in this study, the following will occur:

Your medical records will be looked at and we will ask you questions to make sure you are eligible for the study. You may refuse to answer any question you are asked.

If you are eligible, the study will involve 2 phases lasting up to six months. Phase 1 will take place before you start isotretinoin and Phase 2 will take place while you are receiving isotretinoin.

#### Phase 1 (approximately 4 ½ hours)

For 3 days before the Phase 1 study day, you will be asked to keep track of everything you eat through the smart-phone application "Fooducate" or on a form that we give you. We ask that you not eat grapefruit and not drink grapefruit juice during these 3 days and on your study day.

On the 4<sup>th</sup> day, you will come to the University of Washington for a 4-hour study.

The study will involve you taking a single normal dose of liquid dextromethorphan by mouth. Dextromethorphan is a commonly used cough medication, which is available without a prescription. We will give you water to drink after your dose.

We will ask that you do not eat anything for 4 hours before the start of your study until 1 hour after the start of the study. After that, we will give you a meal. During this fasting time you are encouraged to drink water.

We will measure your height, weight and wrist. We will review your medical record and ask you about medications, vitamins and other things that you are taking as well as your health.

We will have you collect a DNA sample. These are collected by rubbing a brush, like a soft toothbrush, up and down on the inside of each cheek 10 times. We will look at your genes involved in drug handling and response.

We will collect all your urine over 4 hours and a single 2 tablespoons blood sample. These samples will be used to look at genetic material and run tests.

During your study and 1 week after your study, we will ask you questions to find out if you have any problems or complaints.

# Phase 2 (approximately 4 ½ hours)

This study will not affect if you receive isotretinoin or not. Your provider will determine if and how much isotretinoin you need. After you have been on the same dose of isotretinoin for at least 1 week, we will ask that you come in for your Phase 2 study.

The only adjustment in your isotretinoin is that:

- for the 3 days before your phase 2 study, we ask that you take your isotretinoin at the same time everyday,
- you take it at the time that your Phase 2 study day will start and
- you write down the time you take each dose.

We will check to make sure that you can still be in the study by reviewing your medical record and asking you questions.

For 3 days before the Phase 2 study day, you will be asked to keep track of everything you eat through the smart-phone application "Fooducate" or on a form that we give you. We will ask that you not eat grapefruit and not drink grapefruit juice during these 3 days and on your study day.

On the 4<sup>th</sup> day, you will come to the University of Washington for a 4-hour study.

The study will involve you taking a single normal dose of liquid dextromethorphan by mouth. We will give you water to drink after your dose.

We will ask that you do not eat anything for 4 hours before the start of your study until 1 hour after the start of the study. At which time we will give you a meal. During this time, you are encouraged to drink water.

We will measure your height, weight and wrist. We will review your medical record and ask you about medications, vitamins and other things that you are taking as well as your health.

We will collect all your urine over 4 hours and a single 2 tablespoons blood sample. These samples will be used to look at genetic material and run tests.

During your study and 1 week after your study, we will ask you questions to find out if you have any problems or complaints.

All remaining samples at the end of the study will be saved and shared for future research projects.

- I consent to having my leftover samples saved and shared for future research.
- [ ] I do NOT consent to have my leftover samples saved and shared for future research.

## **Study Design Summary**

| | Phase 1 | Phase 2 |
|---|---|---|
| | Prior to Isotretinoin | With Isotretinoin |
| Procedures | Dextromethorphan single dose | Dextromethorphan single dose |
| | 4-hour urine collection | 4-hour urine collection |
| | Single blood sample collection | Single blood sample collection |
| | 3-day food record | 3-day food record |
| | Measure height, weight and wrist | Measure height, weight and wrist |
| | Check for problems or complaints | Check for problems or complaints |
| | DNA collection | 3-day isotretinoin dose record |

The total amount of time for this study is approximately 9 hours. The total amount of blood to be taken for this study will be 4 tablespoons.

## RISKS, STRESS, OR DISCOMFORT

#### **Dextromethorphan Risks:**

Dextromethorphan is often used in children and teenagers. We do not expect that you will have problems with a single dose. However, if you do have problems, the most common will be mild dizziness, sleepiness and tiredness.

Allergic reactions have been reported including rash and rarely anaphylaxis (allergy that causes difficulty breathing).

There may be unanticipated problems from dextromethorphan.

### **Blood Drawing Risks:**

Risks of blood drawing include pain with the needle stick, bruising and rarely fainting or infection. The amount of blood to be drawn for this study will not affect your blood counts.

## **Fasting Risks:**

Risks of not eating for 4 hours before and 1 hour after dextromethorphan dosing include: feeling hungry, gurgling, rumbling or growling in stomach, dizziness, faintness, headache, short-tempered, difficulty paying attention and / or sick to your stomach.

### **Loss of Confidentiality:**

There is a chance when you are in any study that your personal information could be accidently seen by someone not working on the study.

#### Other Risks:

You will receive isotretinoin whether you are in the study or not. Therefore, isotretinoin risks are not risks of this study.

If you have study-related problems or complaints, please contact Dr. Vary through the paging operator at 206-598-6190 and ask for Dr. Vary and call Dr. Hebert at 206-697-2138.

### ALTERNATIVES TO TAKING PART IN THIS STUDY

Taking part in this study is entirely your choice. Choosing not to be in the study will not affect your isotretinoin treatment or your healthcare.

#### BENEFITS OF THE STUDY

There is no direct benefit to you for being in this study. We hope the results of this study will help providers better care for patients needing isotretinoin.

#### SOURCE OF FUNDING

The study team and the University of Washington is receiving financial support for this study from the National Institutes of Health (NIH).

#### CONFIDENTIALITY OF RESEARCH INFORMATION

We will collect personal information such as your name, address, email, phone, date of birth, social security number and medical record number. Coded data will be stored confidentially (linked to identifiers). Coded data will be stored in locked files or on password protected computers. Personal identifiers will not be entered into the computer database.

We have a Certificate of Confidentiality from the federal National Institutes of Health. This helps us protect your privacy. The Certificate means that we do not have to give out identifying information about you even if we are asked to by a court of law. We will use the Certificate to resist any demands for identifying information.

We can't use the Certificate to withhold your research information if you give your written consent to give it to an insurer, employer, or other person. Also, you or a member of your family can share information about yourself or your part in this research if you wish.

There are some limits to this protection. We will voluntarily provide the information to:

- a member of the federal government who needs it in order to audit or evaluate the research;
- individuals at the University of Washington, the funding agency, and other groups involved in the research, if they need the information to make sure the research is being done correctly;
- the federal Food and Drug Administration (FDA), if required by the FDA;
- state or local authorities, if we learn of child abuse, elder abuse, or the intent to harm yourself or others.

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>, as required by U.S. law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

Your participation in this study will be noted in your UW medical record.

There may also be other risks that are not yet known.

## **DATA SHARING**

The National Institutes of Health require that federally funded studies like this study share data with other investigators upon request. If requested, your data will be shared according to the National Institutes of Health requirements. Only coded data will be shared. Your identifying information will not be shared.

#### OTHER INFORMATION

You may refuse to be in and you are free to quit this study at any time without penalty or affect on your healthcare.

You will be paid \$100 for finishing all study procedures associated with each study phase and an additional \$50 for finishing all study procedures. Total payment will be \$250 if all study procedures are completed. Your payment for the study will be less if the study is partially completed. We will need to collect your social security number to pay you.

You will not be charged for any study related procedures.

Printed name of study staff obtaining consent

## **RESEARCH-RELATED INJURY**

Signature

Date

If you think you have a medical problem or illness related to this research, contact Dr. Vary through the paging operator at 206-598-6190 and ask for Dr. Vary and call Dr. Hebert at 206-697-2138 right away. They will treat you or refer you for treatment.

| Subject's sta | atement_ | | |
|---|---|---|---|
| chance to as<br>participating<br>consent form<br>Subjects Div | sk questions. If I hat g in this study, I car m. If I have question vision at (206) 543- | to me. I volunteer to take part in this reve questions later about the research, or contact one of the researchers listed on about my rights as a research subject 0098. I give permission to the research sent form. I will receive a copy of this | or if I have been harmed by<br>on the first page of this<br>ct, I can call the Human<br>hers to use my medical |
| Printed name of subject | | Signature of subject | Date |
| When subje | ct is a minor: | | |
| Printed name of parent | | Signature of parent | Date |
| Copies to: | Researcher<br>Subject<br>Subject's Medic | al Record (if applicable) | |